CLINICAL TRIAL: NCT00253292
Title: Psychometric Study of Outcomes Instruments
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit necessary sample size
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Ronald Tompkins, MD, Sc.D.-PI, Shriners Hospitals for Children
Other Study IDs: 1999-P-008281/15
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Burns; Trauma
Keywords: Burns; Trauma; Outcomes; Quality of Life
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a standardized, practical self-administered questionnaire to monitor young adult burn patients and to evaluate the effectiveness of burn management treatments with regard to improved function, physical appearance and other relevant outcomes.

DETAILED DESCRIPTION:
Identifying young adult burned patients at risk for poor outcomes remains an underpublished field of study. The first step to identifying these patients is to review their responses to this burn specific young adult measure, that attempts to quantify aspects of quality of life. We are validating this questionnaire by now collecting information from non burned community based subjects and by having burned patients complete the questionnaire at 4 timepoints. Once we have recruited sufficient subjects we will finalize our testing of this questionnaire and publish the validity and reliability of the instrument. Our questionnaires will help us answer the question of how burn people differ from non burned person's reported quality of life. This will complete our array of burn specific outcomes questionnaires from infancy through young adulthood.

ELIGIBILITY:
Inclusion Criteria:

* All burn injured young adults with or without grafting
* All burned on or after their 17th birthday
* Between the ages of 19-30
* English speaking
* Present for inpatient or outpatient treatment

Exclusion Criteria:

Non-burned skin conditions

* Non-English speaking
* Patients less than 19 years of age
* Patients over 30 years of age

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients admitted to the MGH burn unit for a burn injury between the ages of 19-30 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 1997-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Tompkins, MD, ScD, Principal Investigator — MGH, Shriners Burn Hospital - Boston
Locations (6):
- United States (6):
  - Shriners Hospital for Children, Sacramento, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jaycee Burn Center,UNC Healthcare, Chapel Hill, North Carolina
  - Shriners Hospitals for Children-Galveston, Galveston, Texas